CLINICAL TRIAL: NCT05180656
Title: The Impact of a Remotely-Delivered Yoga Intervention on Cognitive Function in Breast Cancer Survivors: A Feasibility Study
Brief Title: Feasibility of a Remotely-Delivered Yoga Intervention on Cognitive Function in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Linda Trinh, Professor and Lab Director, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 41494
Record Dates: First submitted 2021-10-04; First posted 2022-01-06 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer; Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will participate in two 60-minute virtual yoga classes each week, delivered through videoconferencing for 8 weeks.
Masking Description: N/A - single-arm study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga Intervention Group (Experimental): All participants will be assigned to the yoga intervention group (single arm).
  Interventions: Behavioral: Yoga Intervention

INTERVENTIONS:
Behavioral: Yoga Intervention — The yoga intervention will consist of two 60-minute yoga classes each week, taught by a certified yoga instructor and delivered remotely through videoconferencing. Participants will be asked to participate in the intervention for 8 weeks.

SUMMARY:
The purpose of this pilot study is to assess the feasibility of a remotely-delivered yoga intervention for breast cancer survivors.

DETAILED DESCRIPTION:
Although up to 75% of breast cancer survivors (BCS) experience cancer-related cognitive impairment (CRCI), there are no proven treatments beyond symptom management. Exercise and yoga interventions for cancer survivors have been shown to be effective in improving other treatment-related side effects such as fatigue, quality of life (QoL), and psychological distress, but there remain several gaps in the exercise oncology literature regarding the optimal type and dose of exercise needed to mitigate CRCI. Specifically, no studies have evaluated the impact of yoga on CRCI using both self-report and objective cognitive measures. Further, no studies have evaluated the impact of a remotely-delivered yoga intervention on CRCI in breast cancer survivors.

Using a mixed-methods approach, this study will will begin to fill these gaps by evaluating the feasibility of a remotely-delivery yoga intervention on cancer-related cognitive impairment (CRCI), fatigue, and exercise levels in individuals diagnosed with breast cancer. The primary objective of this study is to assess the feasibility of a remotely-delivered yoga intervention for breast cancer survivors. This study will inform future randomized controlled trials (RCTs) examining the impact of remotely-delivered yoga interventions, with the eventual goal of providing greater access to exercise programming for symptom management for breast cancer patients and survivors.

All aspects of the study, including the assessments and the yoga intervention will take place remotely through videoconferencing. Feasibility measures, including enrolment, adherence, and attrition rates, as well as adverse events and participant satisfaction, will be tracked and assessed throughout the intervention. Objectively-assessed cognitive function will be measured using the National Institutes of Health (NIH) Virtual Toolbox Cognitive Battery and the online PsyToolkit Task Switching Test. Self-reported cognitive function will be assessed using the Functional Assessment of Cancer Therapy(FACT)-Cognitive questionnaire. Self-reported fatigue will be assessed using the Revised-Piper Fatigue Scale (PFS). Self-reported exercise will be assessed using a modified version of the Godin Leisure Time Exercise questionnaire (GLTEQ). These assessments will be taken at baseline and post-intervention. Participants will be asked to participate in the yoga intervention for 8 weeks. The yoga intervention will consist of two 60-minute yoga classes each week, which will be taught by a certified yoga instructor. Following the intervention, a sub-sample of participants will be will be purposefully selected and asked to participate in semi-structured qualitative interviews to understand their experiences with the intervention and study.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* primary diagnosis of Stage I-IIIa breast cancer
* completed primary treatment(s)
* proficient in written and spoken English
* access to the Internet and a computer with videoconferencing capabilities

Exclusion Criteria:

* colour-blind since the objective cognitive tests require participants to distinguish between colours
* regular yoga practice defined as ≥2 times/week
* major cognitive disorder(s) or impairment(s) (score ≤21 on the Telephone Interview of Cognitive Status)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Enrolment rate | From beginning to end of recruitment period, up to 6 months.
  Participant enrolment rate will be one measure of feasibility. This will be calculated as the number of participants who enrol in the intervention, divided by the total number of participants assessed for study eligibility.
Adherence rate | From beginning to end of intervention period, up to 6 months.
  Adherence rate, or participants' adherence to the intervention, will be one measure of feasibility. This will be calculated as the number of classes participants attend, divided by the number of classes participants are expected to attend throughout the intervention.
Attrition rate | From beginning to end of intervention period, up to 6 months.
  Attrition rate, or participant drop-out, will be one measure of feasibility. This will be calculated as the number of participants who do not complete the intervention, divided by the number of participants enrolled at the post-intervention mark.
Adverse events | From beginning to end of intervention period, up to 6 months.
  Adverse events will be one measure of feasibility. This will be assessed as an unexpected and severe medical problem or injury that occurs during the yoga classes.
Burden and satisfaction | 8 weeks post-baseline
  Burden and satisfaction scores will be one measure of feasibility. This will be assessed using a researcher-generated 15-item questionnaire that asks participants about their experience with the intervention and assessments. Participants will rate items using a 5-point Likert scale (1 = 'strongly disagree', 5 = 'strongly agree').

SECONDARY OUTCOMES:
Self-reported cognitive function | Baseline to 8 weeks post-baseline
  Self-reported cognitive function will be assessed using the 37-item FACT-Cog (Version 3) questionnaire which asks participants about perceived cognitive impairments, comments from others, perceived cognitive abilities, and impact on quality of life. Participants will be asked to rate each item on a 5-point Likert scale (0 = 'never/not at all', 4 = 'several times a day/very much').
Objectively-assessed cognitive function | Baseline to 8 weeks post-baseline
  Objectively-assessed cognitive function will be measured using the National Institutes of Health (NIH) Toolbox Virtual Cognitive battery to measure immediate and working memory, verbal learning, executive function, and language, and the PsyToolkit task switching test to measure executive function. These tests will be administered remotely to participants via an iPad and videoconferencing.
Self-reported fatigue | Baseline to 8 weeks post-baseline
  Self-reported fatigue will be assessed using the Revised-Piper Fatigue Scale questionnaire which is a 27-item questionnaire that asks participants about the degree of their perceived fatigue. Participants will be asked to rate each item on a 10-point Likert scale (0 = 'none', 10 = 'very much')
Self-reported exercise | Baseline to 8 weeks post-baseline
  Self-reported exercise will be assessed using a modified version of the Godin Leisure Time Exercise Questionnaire, which asks participants about the number of times/week and average duration spent in light, moderate, and vigorous exercise in a typical week (7 days) over the past month.
Semi-structured qualitative interviews | 8 weeks post-baseline
  The researcher will conduct semi-structured qualitative interviews over videoconferencing that will ask participants about their experience with the study and intervention, including enjoyment, potential barriers faced, and how they felt physically and cognitively during and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Trinh, PhD, Study Director — University of Toronto, Faculty of Kinesiology and Physical Education
Locations (1):
- Faculty of Kinesiology and Physical Education, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahles TA, Saykin AJ, McDonald BC, Li Y, Furstenberg CT, Hanscom BS, Mulrooney TJ, Schwartz GN, Kaufman PA. Longitudinal assessment of cognitive changes associated with adjuvant treatment for breast cancer: impact of age and cognitive reserve. J Clin Oncol. 2010 Oct 10;28(29):4434-40. doi: 10.1200/JCO.2009.27.0827. Epub 2010 Sep 13. PMID 20837957
- [Background] Bernstein LJ, McCreath GA, Komeylian Z, Rich JB. Cognitive impairment in breast cancer survivors treated with chemotherapy depends on control group type and cognitive domains assessed: A multilevel meta-analysis. Neurosci Biobehav Rev. 2017 Dec;83:417-428. doi: 10.1016/j.neubiorev.2017.10.028. Epub 2017 Oct 29. PMID 29092778
- [Background] Bhattacharyya KK, Andel R, Small BJ. Effects of yoga-related mind-body therapies on cognitive function in older adults: A systematic review with meta-analysis. Arch Gerontol Geriatr. 2021 Mar-Apr;93:104319. doi: 10.1016/j.archger.2020.104319. Epub 2020 Dec 7. PMID 33338831
- [Background] Buffart LM, van Uffelen JG, Riphagen II, Brug J, van Mechelen W, Brown WJ, Chinapaw MJ. Physical and psychosocial benefits of yoga in cancer patients and survivors, a systematic review and meta-analysis of randomized controlled trials. BMC Cancer. 2012 Nov 27;12:559. doi: 10.1186/1471-2407-12-559. PMID 23181734
- [Background] Campbell KL, Zadravec K, Bland KA, Chesley E, Wolf F, Janelsins MC. The Effect of Exercise on Cancer-Related Cognitive Impairment and Applications for Physical Therapy: Systematic Review of Randomized Controlled Trials. Phys Ther. 2020 Mar 10;100(3):523-542. doi: 10.1093/ptj/pzz090. PMID 32065236
- [Background] Carson JW, Carson KM, Porter LS, Keefe FJ, Shaw H, Miller JM. Yoga for women with metastatic breast cancer: results from a pilot study. J Pain Symptom Manage. 2007 Mar;33(3):331-41. doi: 10.1016/j.jpainsymman.2006.08.009. PMID 17349503
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Danhauer SC, Addington EL, Cohen L, Sohl SJ, Van Puymbroeck M, Albinati NK, Culos-Reed SN. Yoga for symptom management in oncology: A review of the evidence base and future directions for research. Cancer. 2019 Jun 15;125(12):1979-1989. doi: 10.1002/cncr.31979. Epub 2019 Apr 1. PMID 30933317
- [Background] Danhauer SC, Griffin LP, Avis NE, Sohl SJ, Jesse MT, Addington EL, Lawrence JA, Messino MJ, Giguere JK, Lucas SL, Wiliford SK, Shaw E. Feasibility of implementing a community-based randomized trial of yoga for women undergoing chemotherapy for breast cancer. J Community Support Oncol. 2015 Apr;13(4):139-147. doi: 10.12788/jcso.0125. PMID 28713846
- [Background] Derry HM, Jaremka LM, Bennett JM, Peng J, Andridge R, Shapiro C, Malarkey WB, Emery CF, Layman R, Mrozek E, Glaser R, Kiecolt-Glaser JK. Yoga and self-reported cognitive problems in breast cancer survivors: a randomized controlled trial. Psychooncology. 2015 Aug;24(8):958-66. doi: 10.1002/pon.3707. Epub 2014 Oct 21. PMID 25336068
- [Background] Eldridge SM, Lancaster GA, Campbell MJ, Thabane L, Hopewell S, Coleman CL, Bond CM. Defining Feasibility and Pilot Studies in Preparation for Randomised Controlled Trials: Development of a Conceptual Framework. PLoS One. 2016 Mar 15;11(3):e0150205. doi: 10.1371/journal.pone.0150205. eCollection 2016. PMID 26978655
- [Background] Galantino ML, Greene L, Daniels L, Dooley B, Muscatello L, O'Donnell L. Longitudinal impact of yoga on chemotherapy-related cognitive impairment and quality of life in women with early stage breast cancer: a case series. Explore (NY). 2012 Mar-Apr;8(2):127-35. doi: 10.1016/j.explore.2011.12.001. PMID 22385567
- [Background] Gothe NP, Kramer AF, McAuley E. The effects of an 8-week Hatha yoga intervention on executive function in older adults. J Gerontol A Biol Sci Med Sci. 2014 Sep;69(9):1109-16. doi: 10.1093/gerona/glu095. Epub 2014 Jul 14. PMID 25024234
- [Background] Janelsins MC, Peppone LJ, Heckler CE, Kesler SR, Sprod LK, Atkins J, Melnik M, Kamen C, Giguere J, Messino MJ, Mohile SG, Mustian KM. YOCAS(c)(R) Yoga Reduces Self-reported Memory Difficulty in Cancer Survivors in a Nationwide Randomized Clinical Trial: Investigating Relationships Between Memory and Sleep. Integr Cancer Ther. 2016 Sep;15(3):263-71. doi: 10.1177/1534735415617021. Epub 2015 Nov 29. PMID 26621521
- [Background] Komatsu H, Yagasaki K, Yamauchi H, Yamauchi T, Takebayashi T. A self-directed home yoga programme for women with breast cancer during chemotherapy: A feasibility study. Int J Nurs Pract. 2016 Jun;22(3):258-66. doi: 10.1111/ijn.12419. Epub 2015 Dec 7. PMID 26643264
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Background] Leon AC, Davis LL, Kraemer HC. The role and interpretation of pilot studies in clinical research. J Psychiatr Res. 2011 May;45(5):626-9. doi: 10.1016/j.jpsychires.2010.10.008. Epub 2010 Oct 28. PMID 21035130
- [Background] Levine AS, Balk JL. Pilot study of yoga for breast cancer survivors with poor quality of life. Complement Ther Clin Pract. 2012 Nov;18(4):241-5. doi: 10.1016/j.ctcp.2012.06.007. Epub 2012 Aug 3. PMID 23059439
- [Background] Newton RU, Hart NH, Clay T. Keeping Patients With Cancer Exercising in the Age of COVID-19. JCO Oncol Pract. 2020 Oct;16(10):656-664. doi: 10.1200/OP.20.00210. Epub 2020 Jun 30. PMID 32603253
- [Background] O'Neill M, Samaroo D, Lopez C, Tomlinson G, Santa Mina D, Sabiston C, Culos-Reed N, Alibhai SMH. The Effect of Yoga Interventions on Cancer-Related Fatigue and Quality of Life for Women with Breast Cancer: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Integr Cancer Ther. 2020 Jan-Dec;19:1534735420959882. doi: 10.1177/1534735420959882. PMID 33073636
- [Background] Ross Zahavich AN, Robinson JA, Paskevich D, Culos-Reed SN. Examining a therapeutic yoga program for prostate cancer survivors. Integr Cancer Ther. 2013 Mar;12(2):113-25. doi: 10.1177/1534735412446862. Epub 2012 Jun 27. PMID 22740082
- [Background] Song, M.-K., Sandelowski, M., & Happ, M. B. (2015). Current practices and emerging trends in conducting mixed methods intervention studies in the health sciences. In A. Tashakkori & C. Teddlie (Eds.), SAGE Handbook of Mixed Methods in Social & Behavioral Research (2nd ed., pp. 725-748). Sage Publications. https://doi.org/10.4135/9781506335193.n28
- [Background] Speed-Andrews AE, Stevinson C, Belanger LJ, Mirus JJ, Courneya KS. Pilot evaluation of an Iyengar yoga program for breast cancer survivors. Cancer Nurs. 2010 Sep-Oct;33(5):369-81. doi: 10.1097/NCC.0b013e3181cfb55a. PMID 20467310
- [Background] Trinh L, Kramer AF, Rowland K, Strom DA, Wong JN, McAuley E. A pilot feasibility randomized controlled trial adding behavioral counseling to supervised physical activity in prostate cancer survivors: behavior change in prostate cancer survivors trial (BOOST). J Behav Med. 2021 Apr;44(2):172-186. doi: 10.1007/s10865-020-00185-8. Epub 2020 Sep 26. PMID 32979134
- [Background] Wefel JS, Vardy J, Ahles T, Schagen SB. International Cognition and Cancer Task Force recommendations to harmonise studies of cognitive function in patients with cancer. Lancet Oncol. 2011 Jul;12(7):703-8. doi: 10.1016/S1470-2045(10)70294-1. Epub 2011 Feb 25. PMID 21354373
- [Background] Yao C, Bernstein LJ, Rich JB. Executive functioning impairment in women treated with chemotherapy for breast cancer: a systematic review. Breast Cancer Res Treat. 2017 Nov;166(1):15-28. doi: 10.1007/s10549-017-4376-4. Epub 2017 Jul 13. PMID 28707202